CLINICAL TRIAL: NCT00003827
Title: Treatment of Poor Risk Myelodysplasia With the Combination of Amifostine, Topotecan and ARA-C: A Phase II Study
Brief Title: Combination Chemotherapy in Treating Patients With Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ALZA (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066982; CHNMC-IRB-98056; ALZA-CHNMC-IRB-98056; NCI-V99-1533
Record Dates: First submitted 1999-11-01; First posted 2003-09-25 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2007-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Amifostine; Cytarabine; Topotecan

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cytarabine
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combining topotecan and cytarabine given with amifostine in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects of amifostine, topotecan, and cytarabine in patients with poor risk myelodysplastic syndrome.
* Determine the hematologic response rate, cytogenetic response rate, and the rate of polyclonal hematopoiesis following this treatment regimen.
* Determine the duration of response and time to disease progression following this treatment regimen in these patients.

OUTLINE: Patients receive topotecan by continuous IV over 24 hours plus cytarabine IV over 2 hours, on days 1-5. Patients receive amifostine IV over 15 minutes every other day for a maximum of 60 days. Patients may receive a second course of the same regimen 8 weeks after the first.

Patients are followed at least monthly for 2 years, then every 3-6 months until death.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study within 1 to 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed poor risk myelodysplastic syndrome, including at least one of the following:

  * Bilineage cytopenia
  * Unfavorable cytogenetic abnormalities
  * Refractory anemia with excess blasts and/or refractory anemia with excess blast in transformation (greater than 5% blast)
* At least 0.5 on the International Prognostic Score System
* No chronic myelomonocytic leukemia
* No hypocellular myelodysplastic syndrome (marrow cellularity less than 30%)

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count less than 1,500/mm3
* Platelet count less than 100,000/mm3
* Hemoglobin less than 10 g/dL

Hepatic:

* ALT less than 5 times upper limit of normal

Renal:

* Creatinine no greater than 1.4 mg/dL

Cardiovascular:

* No congestive heart failure

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Must have right atrial catheter inserted

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior blood or bone marrow transplantations

Chemotherapy:

* No prior acute myeloid leukemia chemotherapy (except hydroxyurea or low dose cytarabine)
* No prior topotecan
* No prior amifostine

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 24 hours since prior antihypertensive medication prior to amifostine

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Fung, MD, FRCPE, Study Chair — City of Hope Comprehensive Cancer Center
Locations (1):
- Cancer Center and Beckman Research Institute, City of Hope, Duarte, California, United States